CLINICAL TRIAL: NCT02472379
Title: Writing About Experiences and Health in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Naomi Eisenberger, Associate Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: GEN; F31AG048668 (NIH); UL1TR000124 (NIH); R03AG049254 (NIH)
Record Dates: First submitted 2015-06-10; First posted 2015-06-15 (Estimated); Last update posted 2017-05-02 (Actual); Status verified 2017-05

CONDITIONS: Social Psychology
Keywords: Immune System; Behavioral Sciences; Women's Health; Health Psychology; Writing

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Writing: Group 1 (Experimental): Subjects will be asked to write about experiences with familiar individuals in their lives.
  Interventions: Behavioral: Writing: Group 1
- Writing: Group 2 (Placebo Comparator): Subjects will be asked to write about experiences with familiar places in their lives.
  Interventions: Other: Writing: Group 2

INTERVENTIONS:
Behavioral: Writing: Group 1 — Writing about experiences with familiar individuals in their lives, once a week for 6 weeks.
  Arms: Writing: Group 1
Other: Writing: Group 2 — Writing about experiences with familiar places, once a week for 6 weeks.
  Arms: Writing: Group 2

SUMMARY:
UCLA researchers looking for healthy females (age 60+) to participate in a study investigating how writing about your experiences may be related to your health.

Once a week for 6 weeks, participants will write about their experiences and fill out online questionnaires. Participants will also come to the UCLA campus for blood draws and to fill out questionnaires 3 times: once prior to the 6-week writing period, once immediately after the 6-week period, and once 2-months after the writing period.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults 60 years and older

Exclusion Criteria:

* Following a structured telephone interview, participants with the following conditions will not be able to participate:

  1. current smokers
  2. active, uncontrolled medical disorders
  3. chronic infection (e.g., Hepatitis C, HIV)
  4. use of certain medications (e.g., hypnotic and psychotropic medication, steroid use, opioid use)
  5. psychiatric disorders (e.g., current major depression, bipolar disorder)
  6. body mass index (BMI) greater than 35

Other exclusion criteria may apply.

Ages: 60 Years to 100 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2015-10; Primary Completion 2017-01 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Inflammatory activity | baseline, post 6-week writing period, 2-months post-writing period
  Changes in proinflammatory cytokine and proinflammatory gene expression from blood draws
Health and well-being (self-report) | baseline, post 6-week writing period, 2-months post-writing period
  Changes in self-report measures of health (e.g., pain, sleep) and well-being (e.g., social support, depression)

CONTACTS AND LOCATIONS:
Overall Officials: Naomi I. Eisenberger, Ph.D., Principal Investigator — University of California, Los Angeles; Mona Moieni, M.A., Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Clinical & Translational Research Center (CTRC), Los Angeles, California, United States